CLINICAL TRIAL: NCT06544538
Title: Causes and Clinical Outcomes of Acute Kidney Injury After Cardiac Arrest: A Retrospective Cohort Study
Brief Title: Acute Kidney Injury After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023/250
Record Dates: First submitted 2024-07-27; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acute Kidney Injury
Keywords: cardiac arrest; Acute kidney injury; Mortality
MeSH Terms: conditions — Acute Kidney Injury; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI Group: AKI 1-3 in the first 48 hours after cardiac arrest according to KDIGO 2012 criteria
- Non-AKI Group: Those who did not develop AKI in the first 48 hours after cardiac arrest according to KDIGO 2012 criteria

SUMMARY:
The development of AKI (Acute Kidney Injury) after cardiac arrest is a common factor associated with mortality. In this study, we aimed to evaluate the factors that increase the risk of developing AKI after cardiac arrest.

For the study, patients were evaluated for the incidence of acute kidney injury (AKI), factors that increase the risk of AKI, and the impact of AKI on mortality. In this process, demographic data, comorbidities, hemodynamic data, laboratory data, clinical symptoms and findings recorded in the electronic decision support system were recorded and analyzed.

DETAILED DESCRIPTION:
This retrospective study was performed on patients hospitalized in intensive care units after cardiac arrest between 2013 and 2022. Patients who met the inclusion criteria were included in the study. Urea, creatinine values, and whether AKI was diagnosed or not were obtained from the data registry system. Statistical evaluation was performed using univariate binary logistic regression analysis.

Demographic data, location of cardiac arrest (in-hospital, out-of-hospital), and duration of CPR were recorded. In addition, the causes of cardiac arrest, HR/MAP (heart rate/average arterial pressure) ratio, and whether VSP (vasopressor) or INO (inotropic) medication was needed were recorded.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with spontaneous circulation after cardiac arrest and admitted to the intensive care unit

Exclusion Criteria:

* Deaths in the first 48 hours
* Missing data
* End stage CKD or first day hemadsorption
* CPR time <3 min
* Unwitnessed cardiac arrest
* Terminal malignancy

  * 90 years old
* Having a pace marker
* Massive bleeding
* ECMO application
* First day diyabetes insipitus

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Anesthesiology and Reanimation intensive care unit of Bakırköy Dr. Sadi Konuk Training and Research Hospital after cardiac arrest
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury (AKI) | Within 48 hours after intensive care unit admission
  Creatinine values in the first 48 hours of intensive care unit admission after cardiac arrest

SECONDARY OUTCOMES:
AKI incidence | Within 48 hours after intensive care unit admission
  Determination of the incidence of AKI development after cardiac arrest
Mortality | Clinical and laboratory data within 48 hours after intensive care unit admission will be used
  Impact of AKI development on mortality in the early post-cardiac arrest period

CONTACTS AND LOCATIONS:
Overall Officials: MURAT ASLAN, Dr, Principal Investigator — Istanbul Bakırköy Dr Sadi Konuk Training and Research Hospital
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data available from the publication date can start If requested, data will be shared with medical doctors dealing with
Supporting Information: Study Protocol, SAP, ICF
Time Frame: to be determined later
Access Criteria: to be determined later

REFERENCES:
- [Background] Nolan JP, Sandroni C, Bottiger BW, Cariou A, Cronberg T, Friberg H, Genbrugge C, Haywood K, Lilja G, Moulaert VRM, Nikolaou N, Olasveengen TM, Skrifvars MB, Taccone F, Soar J. European Resuscitation Council and European Society of Intensive Care Medicine guidelines 2021: post-resuscitation care. Intensive Care Med. 2021 Apr;47(4):369-421. doi: 10.1007/s00134-021-06368-4. Epub 2021 Mar 25. PMID 33765189
- [Background] Kalogeris T, Baines CP, Krenz M, Korthuis RJ. Ischemia/Reperfusion. Compr Physiol. 2016 Dec 6;7(1):113-170. doi: 10.1002/cphy.c160006. PMID 28135002
- [Background] Lemiale V, Dumas F, Mongardon N, Giovanetti O, Charpentier J, Chiche JD, Carli P, Mira JP, Nolan J, Cariou A. Intensive care unit mortality after cardiac arrest: the relative contribution of shock and brain injury in a large cohort. Intensive Care Med. 2013 Nov;39(11):1972-80. doi: 10.1007/s00134-013-3043-4. Epub 2013 Aug 14. PMID 23942856
- [Background] Adler C, Reuter H, Seck C, Hellmich M, Zobel C. Fluid therapy and acute kidney injury in cardiogenic shock after cardiac arrest. Resuscitation. 2013 Feb;84(2):194-9. doi: 10.1016/j.resuscitation.2012.06.013. Epub 2012 Jun 30. PMID 22750662
- [Background] Patyna S, Riekert K, Buettner S, Wagner A, Volk J, Weiler H, Erath-Honold JW, Geiger H, Fichtlscherer S, Honold J. Acute kidney injury after in-hospital cardiac arrest in a predominant internal medicine and cardiology patient population: incidence, risk factors, and impact on survival. Ren Fail. 2021 Dec;43(1):1163-1169. doi: 10.1080/0886022X.2021.1956538. PMID 34315321